CLINICAL TRIAL: NCT00996203
Title: Local Open-label Multicenter Study to Evaluate the Quality of Life in Patients With Moderate to Severe Active Rheumatoid Arthritis and an Inadequate Response to DMARDs When Adding Tocilizumab (TCZ)
Brief Title: A Study of Tocilizumab Added to DMARDs in Patients With Moderate to Severe Rheumatoid Arthritis and an Inadequate Response to DMARDs.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22665
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Antirheumatic Agents

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]; Drug: DMARDs (disease-modifying antirheumatic drugs)

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg iv every 4 weeks for 24 weeks
Drug: DMARDs (disease-modifying antirheumatic drugs) — stable doses at investigator's prescription

SUMMARY:
This open-label single arm study will evaluate the efficacy and safety of tocilizumab added to traditional disease-modifying antirheumatic drugs (DMARDs) in patients with moderate to severe active rheumatoid arthritis and an inadequate response to DMARDs. Patients will receive tocilizumab 8 mg/kg by intravenous infusion every 4 weeks for 24 weeks, in addition to their current non-biologic DMARDs at stable doses. Anticipated time on study treatment is 24 weeks, and the target sample size is 200.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/= 18 years of age
* moderate to severe active rheumatoid arthritis of >/=6 months duration
* inadequate clinical response to current non-biologic DMARDs
* current DMARDs must be at stable dose for 8 weeks prior to study entry
* oral corticosteroids (</=10mg/day prednisone or equivalent) and NSAIDs must be at stable dose for >/=4 weeks prior to screening

Exclusion Criteria:

* rheumatic autoimmune disease other than RA
* history of or current inflammatory joint disease other than RA
* previous treatment with any biologic DMARD
* functional class IV as defined by the ACR classification
* intra-articular or parenteral corticosteroids within 6 weeks prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2009-10-31 (Actual); Primary Completion 2011-02-14 (Actual); Study Completion 2011-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (28):
- Russia (28):
  - Chelyabinsk Regional Clinical Hospital; Rheumatology, Chelyabinsk
  - Republican clinical hospital of Karachai-Cherkess; Rheumatologic Department, Cherkess
  - Irkutsk Regional Consulting and Diagnostic Clinical Center; Regional Center of Reumatolodic Deasise, Irkutsk
  - Republican Clinicodiagnostic Center, Izhevsk
  - Kaliningrad Regional Clinical Hospital; Rheumatologic Department, Kaliningrad
  - War Veterans Regional Clinical Hospital;Therapy Department, Kemerovo
  - Kirov Regional Clinical Hospital; Reumatology Department, Kirov
  - GUZ Regional clinical hospital # 1, Krasnodar
  - GMU Kursk regional clinical hospital, Kursk
  - FSBI "Scientific Research Institute of Rheumatology" of russian Academy of Medical Sciences, Moscow
  - FSBI "FSCC of particularized sorts of medical care and medical technologies of FMBA", Moscow
  - FGU Central Clinical Hospital with Polyclinic Administration President RF, Moscow
  - Head Clinical Hospital of Internal Affair Ministry of Russia, Moscow
  - Vladimirskiy Regional Scientific Research Inst., Moscow
  - SIH Nizhny Novgorod Regional Clinical Hospital n.a. Semashko, Nizhny Novgorod
  - Republican Hospital Named After V.A. Baranov, Petrozavodsk
  - Rostov State Medical University; Cardiorheumatology Department, Rostov-on-Don
  - Clinical hospital #1, Smolensk
  - Surgut Region Clinical Hospital, Surgut
  - Glpu Tjumen Regional Clinical Hospital #1, Tyumen
  - Republican clinical hospital named after G.G. Kuvatov, Ufa
  - State Institution of Healthcare Ulyanovsk Regional Clinical Hospital, Ulyanovsk
  - GUZ "Novgorod Regional Clinical Hospital"; Cardioreumatological, Veliky Novgorod
  - Budget Institution of Healthcare of Voronezh Region "Voronezh Regional Clinical Hospital #1", Voronezh
  - Voronezh Regional Clinical Hospital #1, Voronezh
  - SHI Yaroslavl Regional Clinical Hospital, Yaroslavl
  - Municipal Autonomous Institution of Healthcare "City Clinical Hospital #40", Yekaterinburg
  - Sverdlovsk Regional Clinical Hospital # 1; Rheumatology Dept, Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Participants received tocilizumab 8 milligrams per kilogram (mg/kg) (but not more than 800 mg), intravenously (IV), every 4 weeks for 24 weeks. Participants received a total of 6 infusions.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 201
Completed | 194
Not Completed | 7
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 1
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Population: Safety population: All patients who received at least one dose and had at least one safety assessment after the drug administration.
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg (but not more than 800 mg), IV, every 4 weeks for 24 weeks. Participants received a total of 6 infusions.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Health Assessment Questionnaire (HAQ) Score
Description: HAQ includes 20 questions concerning participant's activities of daily life, grouped in 8 scales of 2 to 3 questions for each activity. To respond to each question, a four-level response (score of 0 to 3 points), with higher scores showing larger functional limitations, was chosen. Scoring was as follows with respect to performance of participant's everyday activities: 0 (equals)=without difficulties; 1=with some difficulties; 2=with great difficulties; and 3=unable to perform these actions at all. Minimum score was 0, maximum score was 3. Withdrawal Visit is the final visit prior to the withdrawal of the subject from the study.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24 and Withdrawal Visit
Population: Intent-to-Treat (ITT) population: All participants randomized in the study who received administration of at least one dose of the study drug and who had at least one efficacy assessment performed. n (number) = number of participants assessed at a specific visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 201
units on a scale
  Week 0 (n=201) | 1.93 (0.60)
  Week 4 (n=199) | 1.49 (0.65)
  Week 8 (n=198) | 1.22 (0.63)
  Week 12 (n=196) | 1.08 (0.62)
  Week 16 (n=193) | 1.00 (0.60)
  Week 20 (n=193) | 0.90 (0.61)
  Week 24 (n=193) | 0.84 (0.62)
  Withdrawal visit (n=6) | 1.32 (1.13)

2. Secondary Outcome: Pain Score as Assessed by Visual Analogue Scale (VAS)
Description: Participant's global assessment of pain was assessed using a 100-millimeter (mm) horizontal VAS (0 to 100 mm) with 0=pain absent and 100=intolerable pain. Participants responded by placing a mark on the line to indicate their current level of pain.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24
Population: ITT Population; n=number of participants assessed at a specific visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 201
mm
  Week 0 (n=201) | 63.82 (16.71)
  Week 4 (n=199) | 46.36 (20.57)
  Week 8 (n=198) | 36.48 (18.94)
  Week 12 (n=196) | 31.90 (19.83)
  Week 16 (n=193) | 26.92 (18.87)
  Week 20 (n=193) | 24.63 (19.09)
  Week 24 (n=193) | 21.96 (18.87)
  Withdrawal visit (n=6) | 34.50 (22.00)

3. Secondary Outcome: European Quality of Life - 5 Dimensions (EQ-5D) Score
Description: EQ-5D questionnaire assess 5 domains of quality of life including mobility, self-care, habitual daily activities, pain, discomfort, and anxiety/depression. Each of five domains was assessed by 3 levels depending on severity of a problem and scored using the following: 1=no disturbances, 2=moderate disturbances, 3=severe disturbances. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24
Population: ITT Population; n=number of participants assessed at a specific visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 200
units on a scale
  Week 0 (n=200) | 0.29 (0.31)
  Week 4 (n=199) | 0.49 (0.24)
  Week 8 (n=198) | 0.57 (0.20)
  Week 12 (n=196) | 0.61 (0.21)
  Week 16 (n=193) | 0.64 (0.19)
  Week 20 (n=193) | 0.66 (0.18)
  Week 24 (n=193) | 0.69 (0.20)
  Withdrawal visit (n=4) | 0.61 (0.07)

4. Secondary Outcome: Change in EQ-5D Score at Week 24 From Baseline
Description: EQ-5D questionnaire assess 5 domains of quality of life including mobility, self-care, habitual daily activities, pain, discomfort, and anxiety/depression. Each of five domains was assessed by 3 levels depending on severity of a problem and scored using the following: 1=no disturbances, 2=moderate disturbances, 3=severe disturbances. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state. Minimum clinically significant change in EQ-5D corresponds to the parameter differences before and after treatment = 0.10. Graduations of assessment of the therapy efficacy by EQ-5D are: Difference (Δ) EQ-5D less than (<)0.10 points: none; 0.10 less than or equal to (≤)Δ EQ-5D ≤0.24: minimal effect; 0.24≤ Δ EQ-5D <0.31: satisfactory effect; Δ EQ-5D greater than or equal to (≥)0.31 points: pronounced effect.
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 200
units on a scale | 0.41 (0.33)
Statistical Analysis 1: Comparison: Tocilizumab; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — EQ-5D scores at Baseline Versus Week 24

5. Secondary Outcome: General Health Score as Assessed by EQ-5D VAS
Description: Participant-reported general health quality was assessed using an EQ-5D 100-mm horizontal VAS (0 to 100 mm) with 0=worst health state and 100=the best health state. The participants were asked to mark the line that corresponded to assessment of general health quality.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24
Population: ITT Population; n=number of participants assessed at a specific visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 201
mm
  Week 0 (n=201) | 39.27 (18.03)
  Week 4 (n=199) | 50.93 (18.78)
  Week 8 (n=198) | 61.79 (43.45)
  Week 12 (n=196) | 66.13 (19.91)
  Week 16 (n=193) | 70.48 (19.39)
  Week 20 (n=192) | 73.31 (19.58)
  Week 24 (n=193) | 76.22 (19.25)
  Withdrawal visit (n=4) | 60.50 (27.77)

6. Secondary Outcome: Percentage of Participants Achieving a Positive Response on Health Quality Assessment of EQ-5D
Description: Participant-reported general health quality was assessed using an EQ-5D 100-mm horizontal VAS (0 to 100 mm) with 0=worst health state and 100=the best health state. The participants were asked to mark the line that corresponded to assessment of general health quality. Positive response was defined as an increase of EQ-5D score by 0.1 or more i.e. it is a clinically significant increase.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24
Population: ITT Population; n=number of participants assessed at a specific visit.
Measure: Number; unit: percentage of Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 198
percentage of Participants
  Week 4 (n=198) | 42.9
  Week 8 (n=198) | 55.6
  Week 12 (n=196) | 60.2
  Week 16 (n=193) | 65.8
  Week 20 (n=193) | 68.4
  Week 24 (n=193) | 73.1

7. Secondary Outcome: Change in General Health Assessed by VAS
Description: as for outcome 5
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 201
mm | 37.3 (25.75)
Statistical Analysis 1: Comparison: Tocilizumab; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — General health at baseline Versus Week 24

8. Secondary Outcome: Disease Activity Score Based on 28-Joint Count (DAS28)
Description: DAS28 calculated from the number of swollen joints and tender joints using the 28-joint count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and global health assessment (participant rated global assessment of disease activity using 10-mm VAS); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24
Population: ITT Population; n=number of participants assessed at a specific visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 199
units on a scale
  Week 0 (n=199) | 6.748 (0.852)
  Week 4 (n=197) | 4.665 (1.227)
  Week 8 (n=196) | 3.777 (1.279)
  Week 12 (n=193) | 3.347 (1.208)
  Week 16 (n=193) | 2.956 (1.230)
  Week 20 (n=192) | 2.762 (1.111)
  Week 24 (n=191) | 2.637 (1.157)

9. Secondary Outcome: Change in DAS28 Score From Baseline to Week 24
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 199
units on a scale | 4.097 (1.289)
Statistical Analysis 1: Comparison: Tocilizumab; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Baseline Versus Week 24 DAS28 scores

10. Primary Outcome: Percentage of Participants With an HAQ Score Decrease of 20 Percent (%), 50%, and 70% During Tocilizumab Treatment
Description: HAQ includes 20 questions concerning participant's activities of daily life, grouped in 8 scales of 2 to 3 questions for each activity. To respond to each question, a four-level response (score of 0 to 3 points), with higher scores showing larger functional limitations, was chosen. Scoring was as follows with respect to performance of participant's everyday activities: 0=without difficulties; 1=with some difficulties; 2=with great difficulties; and 3=unable to perform these actions at all. Minimum score was 0, maximum score was 3.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population:
Measure: Number; unit: percentage of participants
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg (but not more than 800 mg), IV every 4 weeks for 24 weeks. Participants received a total of 6 infusions.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 199
percentage of participants
  Week 4 ≥20% (n=199) | 51.8
  Week 4 ≥50% (n=199) | 15.6
  Week 4 ≥70% (n=199) | 5.0
  Week 8 ≥20% (n=198) | 72.2
  Week 8 ≥50% (n=198) | 28.8
  Week 8 ≥70% (n=198) | 13.6
  Week 12 ≥ 20% (n=196) | 83.7
  Week 12 ≥50% (n=196) | 42.3
  Week 12 ≥70% (n=196) | 18.9
  Week 16 ≥20% (n=193) | 86.5
  Week 16 ≥50% (n=193) | 51.3
  Week 16 ≥70% (n=193) | 21.8
  Week 20 ≥20% (n=193) | 89.6
  Week 20 ≥50% (n=193) | 56.0
  Week 20 ≥70% (n=193) | 34.2
  Week 24 ≥20% (n=193) | 88.1
  Week 24 ≥50% (n=193) | 61.7
  Week 24 ≥70% (n=193) | 38.3

11. Primary Outcome: Change in HAQ Score at Week 24
Description: as for outcome 10
Time Frame: Baseline and Week 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 199
units on a scale | 1.11 (0.66)
Statistical Analysis 1: Comparison: Tocilizumab; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Mean HAQ scores at Baseline Versus Week 24

12. Secondary Outcome: Percentage of Patients With Varied Disease Activity Assessed Using DAS28 During Tocilizumab Treatment
Description: DAS28 calculated from the number of swollen joints and tender joints using the 28-joint count, the ESR mm/hour, and global health assessment (participant rated global assessment of disease activity using 10-mm VAS); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity. Disease activity: 0=remission (DAS28 less than [<] 2.6), I=low (DAS28 less than or equal to [≤]2.6 to <3.2), II=moderate (DAS28=3.2 to 5.1), III=high (DAS28 greater than [>]5.1).
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24
Population: ITT Population; n=number of participants assessed at a specific visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 199
percentage of participants
  Week 0 moderate activity (n=199) | 2.5
  Week 0 high activity (n=199) | 97.5
  Week 4 remission (n=197) | 3.0
  Week 4 low activity (n=197) | 9.6
  Week 4 moderate activity (n=197) | 52.8
  Week 4 high activity (n=197) | 34.5
  Week 8 remission (n=196) | 17.9
  Week 8 low activity (n=196) | 15.3
  Week 8 moderate activity (n=196) | 51.5
  Week 8 high activity (n=196) | 15.3
  Week 12 remission (n=193) | 25.4
  Week 12 low activity (n=193) | 22.8
  Week 12 moderate activity (n=193) | 42.0
  Week 12 high activity (n=193) | 9.8
  Week 16 remission (n=193) | 41.5
  Week 16 low activity (n=193) | 19.2
  Week 16 moderate activity (n=193) | 33.2
  Week 16 high activity (n=193) | 6.2
  Week 20 remission (n=192) | 44.8
  Week 20 low activity (n=192) | 20.8
  Week 20 moderate activity (n=192) | 30.7
  Week 20 high activity (n=192) | 3.6
  Week 24 remission (n=191) | 51.3
  Week 24, low activity (n=191) | 19.4
  Week 20 moderate activity (n=191) | 26.7
  Week 24 high activity (n=191) | 2.6

13. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20), 50% (ACR50), and 70% (ACR70) Response
Description: ACR20/50/70 response: ≥20%, ≥50%, or ≥70% improvement, respectively, in swollen/tender joint count (66 joints assessed for swelling and 68 joints assessed for tenderness) and in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and acute phase response: C-reactive protein (CRP) or ESR.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24
Population: ITT Population; n=number of participants assessed at a specific visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 201
percentage of participants
  ACR20 Week 4 | 50.2
  ACR20 Week 8 | 76.1
  ACR20 Week 12 | 81.1
  ACR20 Week 16 | 89.6
  ACR20 Week 20 | 91.0
  ACR20 Week 24 | 89.1
  ACR50 Week 4 | 9.5
  ACR50 Week 8 | 27.4
  ACR50 Week 12 | 49.3
  ACR50 Week 16 | 61.2
  ACR50 Week 20 | 67.7
  ACR50 Week 24 | 70.6
  ACR70 Week 4 | 3.0
  ACR70 Week 8 | 10.0
  ACR70 Week 12 | 18.4
  ACR70 Week 16 | 26.9
  ACR70 Week 20 | 39.3
  ACR70 Week 24 | 44.3

14. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Response Based on DAS28
Description: The DAS28-based EULAR response criteria were used to measure individual response as no effect, good effect, and moderate effect, depending on the extent of change from baseline and the level of disease activity reached. Good effect: change from baseline >1.2 with DAS28 score ≤3.2; moderate effect: change from baseline >1.2 with DAS28 score 3.2 to 5.1 or change from baseline >0.6 to <1.2 with DAS28 score <3.2; no effect: change from baseline ≤0.6 or change from baseline >0.6 and ≤1.2 with DAS28 score >5.1.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population; n=number of participants assessed at a specific visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 201
percentage of participants
  Week 4, No effect (n=195) | 15.9
  Week 4, Moderate effect (n=195) | 72.3
  Week 4, Good effect (n=195) | 11.8
  Week 8, No effect (n=194) | 5.7
  Week 8, Moderate effect (n=194) | 61.9
  Week 8, Good effect (=194) | 32.5
  Week 12, No effect (n=191) | 4.7
  Week 12, Moderate effect (n=191) | 47.6
  Week 12, Good effect (n=191) | 47.6
  Week 16, No effect (n=191) | 2.1
  Week 16, Moderate effect (n=191) | 37.7
  Week 16, Good effect (n=191) | 60.2
  Week 20, No effect (n=190) | 0.5
  Week 20, Moderate effect (n=190) | 34.2
  Week 20, Good effect (n=190) | 65.3
  Week 24, No effect (n=189) | 1.1
  Week 24, Moderate effect (n=189) | 28.6
  Week 24, Good effect (n=189) | 70.4

15. Secondary Outcome: C-Reactive Protein
Description: CRP (milligrams/Liter) is a mediator of inflammation, acute phase protein.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population; n=number of participants assessed at a specific visit.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Tocilizumab
Number analyzed (Participants) | 200
mg/L
  Week 0 (n=200) | 33.51 (34.86)
  Week 4 (n=198) | 8.67 (15.00)
  Week 8 (n=194) | 7.62 (19.00)
  Week 12 (n=196) | 5.43 (16.69)
  Week 16 (n=191) | 4.66 (13.48)
  Week 20 (n=193) | 4.92 (14.29)
  Week 24 (n=189) | 4.78 (12.94)
  Withdrawal visit (n=6) | 7.00 (0.20)

16. Secondary Outcome: Erythrocyte Sedimentation Rate
Description: ESR (mm/hr) is used to determine the acute phase response.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population; n=number of participants assessed at a specific visit.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Tocilizumab
Number analyzed (Participants) | 201
mm/hr
  Week 0 (n=201) | 53.33 (30.82)
  Week 4 (n=198) | 15.29 (13.77)
  Week 8 (n=197) | 11.97 (14.95)
  Week 12 (n=193) | 10.00 (10.82)
  Week 16 (n=193) | 11.63 (17.99)
  Week 20 (n=193) | 10.71 (13.24)
  Week 24 (n=193) | 10.95 (13.52)
  Withdrawal visit (n=6) | 15.00 (4.00)

ADVERSE EVENTS:
Time Frame: From baseline Visit up to 24 weeks or until withdrawal
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 12/201
Other Adverse Events (participants affected / at risk) | 46/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=201)
Erysipelatous inflammation (Skin and subcutaneous tissue disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cervical myelopathy (Nervous system disorders) | 1
Localized infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Acute pyelonephritis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Hemorrhagic anemia (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
Toxic hepatitis (Hepatobiliary disorders) | 1
Chronic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=201)
Lymphostasis (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Keratitis (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Oral herpes (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 6
Respiratory tract infection viral (Infections and infestations) | 6
Acute tonsillitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Onychomycosis (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Blood pressure increased (Investigations) | 2
Transaminases increased (Investigations) | 8
Alanine aminotransferase increased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Lower limb fracture (Musculoskeletal and connective tissue disorders) | 1
Upper limb fracture (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Pyelonephritis chronic (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin reactions (Skin and subcutaneous tissue disorders) | 1
Tooth extraction (Surgical and medical procedures) | 1
Haemorrhoids (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights